CLINICAL TRIAL: NCT06665568
Title: Keta-Care - Antidepressant and Anxiolytic Effects of Intranasal Ketamine Self-administration in Palliative Care Cancer Patients: an Open-label Feasibility Study
Brief Title: Effects of Intranasal Ketamine on Depression and Anxiety in Palliative Care Cancer Patients
Acronym: Keta-Care
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Keta-Care; KLS-5644-08-2022 (Other Grant/Funding Number: Swiss Cancer League)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Depressive Symptoms Mild to Moderate in Severity; Anxiety; Quality of Life (QOL); Caregiver Burden; Sleep Quality
Keywords: Ketamine; Caregiver burden; Open-label; feasibility; Anxiety; Depression; Palliative Care; Intranasal
MeSH Terms: conditions — Anxiety Disorders; Caregiver Burden; Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Other): Open-label, flexibly-dosed intranasal ketamine hydrochloride
  Interventions: Drug: Intranasal ketamine hydrochloride

INTERVENTIONS:
Drug: Intranasal ketamine hydrochloride — Flexible-dose intranasal ketamine hydrochloride (5 - 50 mg)

SUMMARY:
With progression of cancer, patients and their caregivers experience challenging emotional distress, which can make them feel depressed and very anxious.

Patients with advanced cancer often do not have long to live. However, most antidepressants take a long time to act and cause unwanted side effects. There is hence a need for a fast acting antidepressant with fewer unwanted side effects.

Ketamine is an effective and fast acting antidepressant originating from pain treatment, which has few unwanted side effects. It can be taken by a patient as a nasal spray when it is needed.

The idea of treating depression and anxiety in cancer patients in palliative care with ketamine nasal spray is new. How effective ketamine will be at reducing depression and anxiety in patients is unknown . It is also unknown whether this kind of treatment will be safe and practical for palliative care patients.

This study aims to answer these questions. Patients will be treated with a low dose (5 mg) of ketamine nasal spray and then measure its effectiveness, practicality and safety. Questionnaires will be used to measure these outcomes.

If treating depression and anxiety with ketamine nasal spray proves to be effective, practical and safe, then it could help to improve the quality of life for palliative care patients and reduce the burden of their caregivers.

DETAILED DESCRIPTION:
With progression of cancer, patients, but also their caregivers, are predisposed to experience challenging emotional distress due to their terminal illness, resulting in depression and anxiety. However, the overall limited survival time and often complex medication regimes complicate a timely and tolerable treatment of these symptoms, when time-consuming psychotherapeutic sessions or classic antidepressant medication with side effects are unfavorable.

Ketamine is an effective and fast acting antidepressant originating from pain treatment, which can be administered non-invasively as easy to handle nasal spray. The possibility of using ketamine as needed, and not necessarily daily as classical antidepressants, limits the occurrence of side effects and has the potential to ease symptom burden in patients as well as caregivers in this vulnerable cohort. Yet, the efficacy and feasibility of intranasal ketamine self-administration in palliative care cancer patients has not been investigated to date.

In the open-label feasibility study proposed here, we aim at assessing the safety, feasibility and efficacy for the treatment of depression and anxiety with low-dose (5 mg per stroke) intranasal ketamine in a population of early palliative care cancer patients in an out-patient setting.

If self-administered nasal ketamine proves efficient and safe in this study population of often neglected palliative care patients, an easy to handle, low-cost and fast-acting drug with lower risk for interactions would be available to ease burden and emotional symptom load, and eventually increase quality of life for patients and caregivers.

ELIGIBILITY:
Inclusion Criteria (patients):

* Informed Consent as documented by signature;
* HADS total score of 6 or greater;
* Age 18 years or older;
* Progressive cancer diagnosis (estimated life expectancy 24 months or more)
* Able to attend study visits;
* Ability to speak and understand German;

Exclusion Criteria (patients):

* Clinician assessed cognitive impairment;
* Clinician assessed alcohol or drug abuse;
* Pregnancy or breast-feeding;
* Severe hypertension (greater than 200/120 mmHg);
* Anamnestic mood disorder (major depressive disorder, treatment resistant depression, etc.);
* Suicidality (C-SSRS total score of "low" or less);
* Weight less than 39 kg, greater than 170 kg;
* Angina pectoris or myocardial infarction in the last 6 months;
* Lifetime abuse or dependence on ketamine or phencyclidine;
* Substance abuse or dependence in the 6 months before screen;
* Nasal obstructions or history of nasal surgery.
* Serious health risk caused by increased blood pressure or intracranial pressure:
* Known aneurysmal vascular disease (including intracranial, thoracic or abdominal aortic or peripheral arterial vessels);
* Known history of intracerebral hemorrhage;
* Recent (within 6 weeks) cardiovascular event including myocardial infarction (MI).

Inclusion criteria (caregivers):

* Informed Consent as documented by signature;
* Age 18 years or older;
* Able to attend study visits;
* Ability to speak and understand German.

Exclusion criteria (caregivers):

- None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms assessed by the MADRS | From start of treatment at week 1 (baseline) to the end of treatment at 8 weeks
  Montgomery- Asberg Depression Scale (MADRS), 10 items, higher values indicate increasing symptom burden and total scores range from 0 to 60.

SECONDARY OUTCOMES:
Change in anxiety assessed by the HAM-A questionnaire | From start of treatment at week 1 (baseline) to the end of treatment at 8 weeks
  Hamilton Anxiety Rating Scale (HAM-A), 14 items, higher values indicate increasing symptom burden and total scores range from 0 to 56.
Change in quality of life assessed by the QLQ-C30 questionnaire | From start of treatment at week 1 (baseline) to the end of treatment at 8 weeks
  EORTC Quality of Life Questionnaire (QLQ-C30), 30 items, higher values of questions 1-28 indicate increasing symptom burden / decreasing quality of life and total scores range from 0 to 112. Higher values on the questionnaires final two questions (29, 30) indicate improved health and quality of life. Total scores on these final two questions range from 0 to 14.
Change in sleep quality assessed by the PSQI questionnaire | From start of treatment at week 1 (baseline), at week 4 and at end of treatment at 8 weeks
  Pittsburgh Sleep Quality Index (PSQI), 10 items, higher values indicate decreasing sleep quality and total scores range from 0 to 21.
Change in depressive symptoms assessed by the HADS questionnaire | From start of treatment at week 1 (baseline) to the end of treatment at 8 weeks
  Hospital Anxiety and Depression Scale (HADS), 14 items, higher values indicate increasing symptom burden and total scores range from 0 to 21.
Change in caregiver burden assessed by the ZBS questionnaire (caregivers) | From start of treatment at week 1 (baseline) to the end of treatment at 8 weeks
  Zarit Burden Scale (ZBS), 22 items, higher values indicate increasing caregiver burden and scores range from 0 to 88.
Change in caregiver quality of life assessed by the CarGoQoL questionnaire (caregivers) | From start of treatment at week 1 (baseline), at week 4 and at end of treatment at 8 weeks
  The CareGiver Oncology Quality of Life Questionnaire (CarGoQoL), 29 items, higher values indicate increasing caregiver quality of life and total scores range from 0 to 100.
Change in sleep quality assessed by the PSQI questionnaire (caregivers) | From start of treatment at week 1 (baseline), at week 4 and at end of treatment at 8 weeks
  Pittsburgh Sleep Quality Index (PSQI), 10 items, higher values indicate decreasing sleep quality and total scores range from 0 to 21.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
We are not required to provide information about plans to share individual participant data (IPD).